CLINICAL TRIAL: NCT03935854
Title: Impact of A Low-Carbohydrate, High-Fat, Ketogenic Diet on Obesity, Metabolic Abnormalities and Psychiatric Symptoms in Patients With Bipolar or Schizophrenia Illness: A Pilot Trial
Brief Title: Impact of a Ketogenic Diet on Metabolic and Psychiatric Health in Patients With Bipolar or Schizophrenia Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shebani Sethi, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48527
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Ketogenic Dieting; Metabolic Syndrome; Bipolar Disorder; Schizophrenia; Weight Gain; Psychotropic Agents Causing Adverse Effects in Therapeutic Use; Brain Metabolic Disorder
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Bipolar Disorder; Schizophrenia; Weight Gain; Brain Diseases, Metabolic | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet 16 Week Group (Experimental): Patients follow ketogenic diet for 16 weeks, with monitoring of physical and psychological health and coaching support
  Interventions: Other: LCHF, Ketogenic Diet

INTERVENTIONS:
Other: LCHF, Ketogenic Diet — Low Carbohydrate, Moderate Protein, High Fat Ketogenic Dietary Intervention 16 weeks

SUMMARY:
To initiate a low-carbohydrate, high-fat (LCHF) or ketogenic dietary (KD) intervention among a cohort of outpatients with either schizophrenia or bipolar illness who also have metabolic abnormalities, overweight/obesity, and/or are currently taking psychotropic medications experiencing metabolic side effects.

DETAILED DESCRIPTION:
Adults with mental illness represent a high-risk, marginalized group in the current metabolic and obesity epidemic. Among US adults with severe mental illness, metabolic syndrome are highly prevalent conditions having severe consequences, with patients estimated to die on average 25 years earlier than the general population largely of premature cardiovascular disease. Many psychiatric medications, particularly neuroleptics and mood stabilizers, may, in addition, contribute to metabolic side effects and weight gain. Low-carbohydrate high-fat (LCHF) or ketogenic diets (KD) have been shown to reduce cardiovascular risk in those with insulin resistance. Recent findings support the idea that bipolar disorder, along with other psychiatric diseases schizophrenia, may have roots of metabolic dysfunction: cerebral glucose hypometabolism, oxidative stress, as well as mitochondrial and neurotransmitter dysfunction which has downstream effects on synapse connections. A KD diet provides alternative fuel to the brain aside from glucose and is believed to contain beneficial neuroprotective effects, including stabilization of brain networks, reduction of inflammation and oxidative stress. The purpose of this study is to evaluate both the metabolic and psychiatric outcomes with a KD diet in this psychiatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Meet DSM V criteria for schizophrenia or bipolar disorder, any subtype, for > 1 year and clinically stable (with no hospitalization for past 3 months)
3. Currently taking psychotropic medication and gained at least 5% weight since starting medication or have a BMI greater than or equal to 26 kg/m2 or presence of at least one metabolic abnormality (hypertriglyceridemia, insulin resistance, dyslipidemia, impaired glucose tolerance)
4. Willing to consent to all study procedures and attend follow-up appointments and motivated to follow the dietary program.
5. Sufficient control over their food intake to adhere to study diets.
6. Willingness to regularly monitor blood pressure, glucose, dietary intake, and body weight over the 4-month trial

Exclusion Criteria:

1. Any subject pregnant or nursing
2. Comorbidity of developmental delay
3. Active substance abuse with illicit drugs or alcohol
4. In a current severe mood or psychotic state when entering the study that would prohibit compliance with study visits or dietary program.
5. Anyone who has been hospitalized or taken clozapine over the past 3 months
6. Inability to complete baseline measurements
7. Severe renal or hepatic insufficiency
8. Cardiovascular dysfunction, including diagnosis of:

   1. Congestive heart failure
   2. Angina
   3. Arrhythmias
   4. Cardiomyopathy
   5. Valvular heart disease
9. Any other medical condition that may make either diet dangerous as determined by the study medical team (e.g. anorexia nervosa)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Change in heart rate from baseline | Baseline, 16 weeks
  Heart rate recorded at 9 visits during study
Change in blood pressure from baseline | Baseline, 16 weeks
  Blood pressure recorded at 9 visits during study
Change in weight from baseline | Baseline, 16 weeks
  Weight recorded at 9 visits during study
Change in waist circumference from baseline | Baseline, 16 weeks
  waist circumference measured at 9 visits during study
Change in visceral fat mass from baseline | Baseline, 16 weeks
  Body composition (SECA) recorded at 5 visits during study
Change in body fat mass from baseline | Baseline, 16 weeks
  Body composition (SECA) recorded at 5 visits during study
Percent Change in Hemoglobin A1c from baseline | Baseline, 16 weeks
  Hemoglobin A1c recorded at initial and final visits
Change in insulin resistance measure (HOMA-IR) from baseline | Baseline, 16 weeks
  HOMA-IR measured at initial and final visits
Change in inflammatory marker (hsCRP) from baseline | Baseline, 16 weeks
  hsCRP measured at initial and final visits
Change in lipid profile TG (triglycerides) from baseline | Baseline, 16 weeks
  Lipid profile TG measured at initial and final visits
Change in lipid profile small LDL (small dense LDL) from baseline | Baseline, 16 weeks
  Lipid profile small LDL measured at initial and final visits
Change in lipid profile (HDL) from baseline | Baseline,16 weeks
  Lipid profile HDL measured at initial and final visits

SECONDARY OUTCOMES:
Psychiatric Indices - Mood | Baseline, 16 weeks
  Change in Mood Qualitative Score (Clinical Mood Monitoring) from baseline
Psychiatric Indices- Clinical Global Impression | Baseline, 16 weeks
  Change in Clinical Global Impression Scales (CGI) from baseline 1-7 scale. 1= not at all ill, 7= among the most extremely ill patients)
Generalized Anxiety Disorder - GAD-7 Anxiety | Baseline, 16 weeks
  Change in Generalized Anxiety Symptom (GAD-7) scale from baseline. 0-15+ scale. (0= no anxiety, 15+= severe anxiety)
Patient Health Questionnaire - PHQ-9 Depression | Baseline, 16 weeks
  Change in Patient Health Questionnaire (PHQ-9) from baseline. Score range 0-27 (0= no depression, 27= severe depression)
Psychiatric Indices- Global Assessment of Functioning | Baseline, 16 weeks
  Change in Global Assessment of Functioning (GAF) Scale from baseline. 1-100 scale (1= persistent danger of hurting self or others, 100= superior functioning)
Psychiatric Indices- Quality of Life | Baseline, 16 weeks
  Change in Manchester Quality of Life Scale (MANSA) from baseline. Range 12-84 (each of 12 outcomes rated from 1= could not be worse to 7= could not be better; <4= dissatisfied with QoL, >4= satisfied with QoL)
Psychiatric Indices- BPRS | Baseline, 16 weeks
  Change in Brief Psychiatric Rating Scale (BPRS) from baseline. Score range 18-126. (For each of 18 symptoms, 1=symptom not present, 7= extremely severe)
Pittsburgh Sleep Quality Index - PSQI | Baseline, 16 weeks
  Change in Pittsburgh Sleep Quality Index from baseline. 0-21 scale (<5=good sleeper; 5+= meaningfully disturbed sleep or poor sleeper)

CONTACTS AND LOCATIONS:
Overall Officials: Shebani Sethi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Psychiatry & Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sethi S, Sinha A, Gearhardt AN. Low carbohydrate ketogenic therapy as a metabolic treatment for binge eating and ultraprocessed food addiction. Curr Opin Endocrinol Diabetes Obes. 2020 Oct;27(5):275-282. doi: 10.1097/MED.0000000000000571. PMID 32773576
- [Background] Carmen M, Safer DL, Saslow LR, Kalayjian T, Mason AE, Westman EC, Sethi S. Treating binge eating and food addiction symptoms with low-carbohydrate Ketogenic diets: a case series. J Eat Disord. 2020 Jan 29;8:2. doi: 10.1186/s40337-020-0278-7. eCollection 2020. PMID 32010444
- [Background] Norwitz NG, Sethi S, Palmer CM. Ketogenic diet as a metabolic treatment for mental illness. Curr Opin Endocrinol Diabetes Obes. 2020 Oct;27(5):269-274. doi: 10.1097/MED.0000000000000564. PMID 32773571
- [Background] Yu B, Ozveren R, Sethi Dalai S. Ketogenic diet as a metabolic therapy for bipolar disorder: Clinical developments. Submitted to Journal of Affective Disorders. Research Square preprint March 2020: DOI is: 10.21203/rs.3.rs-334453/v1
- [Background] Brietzke E, Mansur RB, Subramaniapillai M, Balanza-Martinez V, Vinberg M, Gonzalez-Pinto A, Rosenblat JD, Ho R, McIntyre RS. Ketogenic diet as a metabolic therapy for mood disorders: Evidence and developments. Neurosci Biobehav Rev. 2018 Nov;94:11-16. doi: 10.1016/j.neubiorev.2018.07.020. Epub 2018 Jul 31. PMID 30075165
- [Background] Sarnyai Z, Kraeuter AK, Palmer CM. Ketogenic diet for schizophrenia: clinical implication. Curr Opin Psychiatry. 2019 Sep;32(5):394-401. doi: 10.1097/YCO.0000000000000535. PMID 31192814
- [Result] Sethi S, Wakeham D, Ketter T, Hooshmand F, Bjornstad J, Richards B, Westman E, Krauss RM, Saslow L. Ketogenic Diet Intervention on Metabolic and Psychiatric Health in Bipolar and Schizophrenia: A Pilot Trial. Psychiatry Res. 2024 May;335:115866. doi: 10.1016/j.psychres.2024.115866. Epub 2024 Mar 20. PMID 38547601

DOCUMENTS (1):
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03935854/ICF_000.pdf